CLINICAL TRIAL: NCT02094209
Title: Clinical Data Collection With a Novel Biofeedback Technology for Continuous Monitoring of Bone Healing
Brief Title: Focused Registry SmartFix
Acronym: FRSmartFix
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FRSmartFix
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2018-01

CONDITIONS: Fracture of Shaft of Tibia
Keywords: External Fixation; Tibial fracture; Fracture healing
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SmartFix — AO Fracture Monitor attached postoperatively to a connection rod of the external fixator. The device continuously measures deformation of the fixator frame due to weight bearing for up to 4 months by means of a strain gauge.

SUMMARY:
20 patients having received an AO large external fixator at the tibia will be equipped with a data logger device (AO Fracture Monitor) attached post-operation to a connection rod of the external fixator. The device continuously measures deformation of the fixator frame due to weight bearing for up to 6 months by means of a strain gauge. Several parameters are calculated from the recorded change in the strain signal and are stored at a regular interval.

DETAILED DESCRIPTION:
Maturation of fracture callus leads to unloading of the fracture fixation hardware due to an increased load-share of the repair tissue. A novel data logger device (AO Fracture Monitor) continuously measures the decline in fixation hardware deflection under physiological loading as indirect indicator for the healing progress. Parameters obtained from the data logger device carry potential to significantly improve the assessment of fracture healing in the future. Meaningful interpretation of measurements requires a set of clinical reference data.

20 patients having received an AO large external fixator at the tibia will be equipped with a data logger device (AO Fracture Monitor) attached post-operation to a connection rod of the external fixator. The device continuously measures deformation of the fixator frame due to weight bearing for up to 4 months by means of a strain gauge. Several parameters are calculated from the recorded change in the strain signal and are stored at a regular interval. Data is collected from the AO Fracture Monitor at follow-up visits of the patient by wireless data transfer. Together with additional variables such as treatment details, fracture healing and pain reported by the patient, the collected data is used to build up a database. Data from the AO Fracture Monitor will be correlated with patient data to investigate the relevance and reliability of the data derived from the AO Fracture Monitor.

In this phase, the study does not imply changes on the operational treatment, nor does it allow for therapeutic consequences based on the derived data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of Femoral or tibial fracture (AO 41-43)
* External fracture fixation with AO large external fixator
* Capable of at least partial weight-bearing
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/Informed Consent Form (ICF)
  * Willingness and ability to participate in the Focused Registry according to the Registry Plan (RP)
  * Signed and dated Ethics Committee (EC) approved written informed consent

Exclusion Criteria:

Preoperative exclusion criteria:

* External fixation as temporary stabilization
* Joint-bridging external fixation
* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or nursing mother
* Emergency patient
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Tibia shaft fracture and external fracture fixation (AO large external fixator).
  Patients capable of at least partial weight-bearing (or expected to do so in the course of healing).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in Parameters derived from the AO Fracture Monitor during bone healing | Discharge, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  AO Fracture Monitor:
  * Mean deformation amplitude per 6 hours
  * Mean deformation rate
  * Number of load-cycles
  * Histogram of patient activity (load intensity distribution)

SECONDARY OUTCOMES:
Change in Pain during bone healing | Preoperative, Discharge, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months (after surgery)
  Pain measured with visual analog scale (VAS)
Change in weight-bearing during bone healing | Discharge, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months (after surgery)
  Documentation of allowed weight-bearing
Repeated reference deformation at a load of 20 / 30 kg | Discharge, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months (after surgery)
  Two reference deformation values are measured under a load 20 kg and 30 kg respectively. The patient steps with his injured leg on a bathroom scale and loads it first with the reference load of 20 kg. The investigator then starts the measurement of the corresponding deformation value. After an acoustic signal indicates the end of the measurement, the procedure is repeated with a reference load of 30 kg. If the patient is not able to put the required load on his leg (e.g. due to pain), the reference value should be measured at a lower load with a note of the actually applied load in the patient record.
Patient information | Up to 4 weeks before surgery
  * Patient demographics
  * Comorbidities
Treatment information | Discharge
  * Fracture classification according to AO and Gustilo
  * Reason for external fixator treatment
  * Previous treatment related to current injury, if any
  * Fixator configuration
Development of the radiological healing assessment: RUST system | Discharge, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months (after surgery)
  The Radiographic Union Score for Tibial fractures (RUST score) is a reliable score to assess the healing of tibial fractures. Each of the four cortices (anterior, posterior, medial and lateral) is given a value from 1 to 3, depending on the presence of a callus and the visibility of the fracture line. The sum of the individual cortical scores results in a RUST value between 4 (definitely not healed) to 12 (definitely healed).
  To investigate, whether patient activity as measured by the AO Fracture Monitor correlate with the radiological assessed course of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Dankward Höntzsch, Professor, Principal Investigator — Berufsgenossenschaftliche Unfallklinik Tübingen
Locations (1):
- Berufsgenossenschaftliche Unfallklinik, Tübingen, Baden-Wurttemberg, Germany